CLINICAL TRIAL: NCT05519813
Title: Effects of Pioglitazone Combined With Metformin and Metformin on Gonadal and Metabolic Profiles in Chinese Nonobese PCOS Patients With Hyperandrogenemia.
Brief Title: Effects of Pioglitazone Combined With Metformin on Gonadal and Metabolic Profiles in Chinese Nonobese PCOS Patients.
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Bing He (Other)
Responsible Party: Sponsor-Investigator, Bing He, Professor, Shengjing Hospital
Organization: Shengjing Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: M0741
Record Dates: First submitted 2022-04-13; First posted 2022-08-29 (Actual); Last update posted 2022-08-29 (Actual); Status verified 2022-08

CONDITIONS: Polycystic Ovary Syndrome
MeSH Terms: conditions — Polycystic Ovary Syndrome | interventions — Metformin; Pioglitazone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Use Metformin for 3 months to treat PCOS (Experimental): Active Comparator: Metformin (BMI<24) Subjects: PCOS patients whoseBMI<24 Drug: Glucophage Generic name: Metformin Dosage form: 500mg Dosage: 1500-2000mg/day Frequency: 500mg three times a day/1000mg twice a day Duration: 3 months
  Interventions: Drug: Metformin
- Use Pioglitazone Hydrochloride And Metformin Hydrochloride Tablets for 3 months to treat PCOS (Experimental): Active Comparator: Pioglitazone Hydrochloride And Metformin Hydrochloride Tablets (BMI<24) Subjects: PCOS patients whoseBMI<24 Drug: Pioglitazone Hydrochloride And Metformin Hydrochloride Tablets Generic name: Pioglitazone Hydrochloride And Metformin Hydrochloride Tablets Dosage form: 15mg/500mg Dosage: 2 tablets/day Frequency: one tablet twice a day Duration: 3 months
  Interventions: Drug: Pioglitazone Hydrochloride And Metformin Hydrochloride Tablets

INTERVENTIONS:
Drug: Metformin — Use Metformin for 3 months to treat PCOS
  Arms: Use Metformin for 3 months to treat PCOS
Drug: Pioglitazone Hydrochloride And Metformin Hydrochloride Tablets — Use Pioglitazone Hydrochloride And Metformin Hydrochloride Tablets for 3 months to treat PCOS
  Arms: Use Pioglitazone Hydrochloride And Metformin Hydrochloride Tablets for 3 months to treat PCOS

SUMMARY:
To study the effects of pioglitazone combined with metformin and metformin on gonadal and metabolic profiles in PCOS patients with BMI < 24 in China. 60 cases of nonobese PCOS patients were collected from Shengjing hospital. The intervention period was 3 months after intervention with met or met + ph. To evaluate the improvement of met or met + ph in the treatment of hyperandremia, glucose metabolism, BMI, waist circumference, menstruation, hairiness and acne in PCOS patients.

ELIGIBILITY:
Inclusion Criteria:

1. Females 18 years to 40 years of age Diagnosed as PCOS by the 2003 Rotterdam criteria
2. BMI<24 kg/m2
3. No pregnant plan in recent 6 months
4. Written consent for participation in the study

Exclusion Criteria:

1. type 1 or type 2 diabetes mellitus
2. Subjects have other endocrine diseases, such as adrenal hyperplasias or tumor, androgen-secreting tumors, Cushing's syndrome, thyroid diseases, and hyperprolactinemia
3. Diagnosed with or have a family history of medullary thyroid carcinoma (MTC) or Multiple Endocrine Neoplasia syndrome type 2 (MEN 2)
4. Serious systemic disease or malignant tumor
5. History of pancreatitis (chronic, acute or recurrent)
6. Body weight change ≥10% at 3 months before treatment
7. Used oral contraceptives or sex hormone drugs in the past 1 month
8. Used oral glucocorticoids in the past 1 month
9. Substance (alcohol or drug) abuse or dependence within 3 months
10. Heavy smokers (smokers who smoke 20 or more cigarettes a day) or heavy drinkers (>10g/d)
11. Subjects have a severe systemic disease, such as cardiovascular system, Renal impairment (eGFR<60ml/min/1.73m2)
12. Increase of transaminases up to < 2.5 times of upper limit of normal value
13. Have a history of thromboembolic disease or thrombotic tendency
14. Subjects in pregnant or lactating or within 1 year after delivery
15. Subjects have an allergic history to the drugs used in the study
16. Subjects have participated in other clinical researches of medicine within

    1 month prior to randomization
17. Use of metformin, pioglitazone, or pioglitazone combined with metformin within 30 days before screening

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 60 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2023-01-01 (Estimated); Study Completion 2023-03-20 (Estimated)

PRIMARY OUTCOMES:
Changes in sex hormone binding globulin (SHBG) | 12 weeks
  Changes in sex hormone binding globulin (SHBG)

SECONDARY OUTCOMES:
Changes in free testosterone (FT) | 12 weeks
  Changes in free testosterone (FT)
Changes in Luteinizing Hormone (LH) | 12 weeks
  Changes in Luteinizing Hormone (LH)
Changes in follicle stimulating hormone (FSH) | 12 weeks
  Changes in follicle stimulating hormone (FSH)
Changes in total testosterone (TT) | 12 weeks
  Changes in total testosterone (TT)
Changes in dehydroepiandrosterone sulfate (DHEAS) | 12 weeks
  Changes in dehydroepiandrosterone sulfate (DHEAS)
Changes in anti-müllerian hormone (AMH) | 12 weeks
  Changes in anti-müllerian hormone (AMH)
Changes in progesterone (Prog) | 12 weeks
  Changes in progesterone (Prog)
Changes in prolactin (PRL) | 12 weeks
  Changes in prolactin (PRL)
Changes in Blood Glucose and Insulin During the oral glucose tolerance test (OGTT) | 12 weeks
  glucose obtained at 0 minutes during the OGTT.
Changes in frequency of menstrual cycle | 12 weeks
  Changes in frequency of menstrual cycle
Change in Acne severity score | 12 weeks
  Change in Acne severity score,the range of acne severity score is 0-9, higher scores mean a worse outcome.
Change in Ferriman-Gallwey score | 12 weeks
  Change in Ferriman-Gallwey score#the range of Ferriman-Gallwey score is 0-9, higher scores mean a worse outcome.
Change in waist circumference(WC) | 12 weeks
  Change in waist circumference(WC)

CONTACTS AND LOCATIONS:
Locations (1):
- Shengjing Hospital of China Medical University, Shenyang, Liaoning, China